CLINICAL TRIAL: NCT01620632
Title: Prospective Evaluation of the Clinical Utility of Laparoscopy-assisted ERCP in Patients With Altered Gastric Anatomy
Brief Title: Laparoscopy-assisted ERCP in Patients With Altered Gastric Anatome
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201600462; 511-2011 (Other: UF IRB)
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Biliary Disease; Pancreas Disease
Keywords: laparoscopy assisted ERCP; altered gastric anatomy
MeSH Terms: conditions — Gallbladder Diseases; Pancreatic Diseases | interventions — Cholangiopancreatography, Endoscopic Retrograde; Laparoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Altered gastric anatomy: Patients who have an altered gastric who need an ERCP
  Interventions: Procedure: Laparoscopy assisted ERCP

INTERVENTIONS:
Procedure: Laparoscopy assisted ERCP — Patients will go the the Operating room and through laparoscopy will have an ERCP for their medical indication.
  Other Names: Endoscopic Retrograde Cholangiopancreatography (ERCP); Roux-en-Y gastric bypass surgery; Laparoscopy

SUMMARY:
The purpose of this research study is to collect data on the technical aspects of Lasparoscopy-assisted ERCP and patient outcomes to help guide future medical care of patients with Roux-en-Y gastric bypass surgery.

DETAILED DESCRIPTION:
Patients would have had a Roux-en-Y gastric bypass in the past that had altered their gastric anatomy. Now they have developed bilary and/or pancreatic problems that require and ERCP. With their altered gastric anatomy a standard ERCP would not be possible. Thus they are scheduled for a Laparoscopy-assisted ERCP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Altered gastric anatomy
* Scheduled to undergo laparoscopy-assisted ERCP

Exclusion Criteria:

* Any contraindications to performing endoscopy
* Participation in another research protocol that could interfere or influence the outcomes measures of the present study.
* The subject is unable/unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those patients who have altered gastric anatomy that require a laparoscopy assisted ERCP
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2011-12; Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
patients with altered gastric anatomy who need an ERCP | approximately one week

CONTACTS AND LOCATIONS:
Overall Officials: Peter V Draganov, MD, Principal Investigator — University of Florida
Locations (1):
- Shands at the University of Florida, Gainesville, Florida, United States